CLINICAL TRIAL: NCT07185100
Title: A Prospective, Cross-sectional, Nationwide Community-based Observational Study to Determine the Prevalence of Unrecognized Heart Failure Among Patients at Risk in Urban Areas Across Germany Using CMR
Brief Title: Determination of the Prevalence of Unrecognized Heart Failure Among Patients at Risk in Urban Areas Across Germany Using CMR
Acronym: WE-CARE-HF-CMR
Status: Recruiting | Type: Observational
Sponsor: German Heart Institute (Other)
Collaborators: Medical Statistics, University Medicine of Goettingen (Other); AstraZeneca (Industry)
Responsible Party: Principal Investigator, Sebastian Kelle, Dr. Sebastian Kelle (MD), German Heart Institute
Other Study IDs: WE-CARE-HF-CMR
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure With Preserved Ejection Fraction (HFPEF)
Keywords: Prevention; Heart failure; HFpEF; Asymptomatic; Cardiology; Urban area; Germany; CMR; Cardiac Magnetic Resonance; HFrEF; Diastolic Dysfunction; Strain
MeSH Terms: conditions — Heart Failure; Sprains and Strains

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at risk of heart failure: asymptomatic individuals, residing in urban areas in Germany, between the age of 40 to 69 years without known HF and at least one established cardiovascular risk factor

SUMMARY:
Heart failure (HF) in patients at risk is often overlooked, and when detected, there is a lack of early and effective preventive interventions. The WE-CARE-HF-CMR study, conducted in large cities/metropol areas in Germany ( > 500.000 inhabitants), aims to close this gap by evaluating the feasibility of a mobile, telemedicinemonitored HF-screening approach combining cardiac magnetic resonance imaging (CMR), quality of life assessment and laboratory tests as key elements in asymptomatic patients at risk. WE-CARE-HF-CMR will provide a proposal for a comprehensive, contemporary screening approach for patients at risk to develop HF tailored to the needs of the target population. This will provide important new information on the prevalence of asymptomatic HF in at-risk patients in urban versus rural areas.

The results of the study will be compared with the results from the "HERZCheck'' trial, which provides data from approximately 4,500 participants in rural areas in Germany and has already been completed (NCT05122793).

DETAILED DESCRIPTION:
The WE-CARE-HF-CMR-study is a cross-sectional, nationwide prospective, community-based observational study to improve the diagnosis of heart failure in urban populations with characteristic risk factors for the occurrence of heart failure using telemedically-supervised mobile diagnostic units. The central diagnostic methods employed in the assessed screening routine comprise a questionnaire-based medical history, laboratory testing and a standardized, non-invasive imaging examination.

Within the framework of the study, 450 subjects aged 40 to 69 years and of male, female or diverse gender, who have characteristic risk factors for the occurrence of asymptomatic heart failure will be examined.

The central diagnostic imaging method of the study is a standardized, needle- as well as stress- and contrast-agent-free CMR exam. The examinations are carried out in mobile MRI diagnostic units at various clinic locations in 5 major cities (> 500.000 residents) in Germany. The various clinics were recommended as locations because they offer good infrastructural conditions for setting up the mobile MRI diagnostic units, which are 27 t truck units, and because emergency medical care for the study participants can also be guaranteed. The medical staff of the clinics is not involved in the study. The potential study participants will be informed exclusively via telemedicine by the investigators of the DHZC in a video call either in a room rented specifically for this purpose or in an accompanying vehicle of the mobile MRI diagnostic unit. The consent of the study participants is also obtained via telemedicine and in accordance with current legal requirements in Germany. The planned examinations in the mobile diagnostic unit will be carried out exclusively by the staff of the company operating the MRI units on behalf of and under the telemedical supervision of the investigators and the study management of the DHZC, acting as the central unit.

ELIGIBILITY:
Inclusion Criteria:

Asymptomatic subjects with:

* chronic diabetes mellitus (known/diagnosed and/or antidiabetic medication and/or elevated HbA1C) and/or
* renal impairment (known/diagnosed CKD and/or in laboratory CKD III° or higher) and/or
* Hypertension (known/diagnosed and/or antihypertensive medication/treatment) and/or
* Hypercholesterolaemia (known/diagnosed and/or antilipid medication/treatment) and/or
* Obesity (known/diagnosed and/or BMI > 30 (kg/m²)) and/or
* Smoker (known/diagnosed and/or current/previous and/or medication/treatment)
* Age 40-69 years
* female or male or diverse sex
* Ability to provide informed consent
* Provision of Informed Consent

Exclusion Criteria:

* Inability to provide written informed consent
* Diagnosed heart failure or previously detected reduced ejection fraction
* General MRI exclusion criteria (pacemaker, defibrillator, intracranial aneurysm clips, metallic foreign bodies in the eyes)
* Any MRI exclusion criteria not listed here, as determined by the MRI laboratory performing the procedure
* Haemodynamically unstable participants (heart rate < 45/min, systolic blood pressure < 90 mmHg)
* Claustrophobia
* Sensorineural hearing loss of 30 dB or more and tinnitus
* Acute mental disorders requiring therapy
* In the presence of pregnancy

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population from which the groups or cohorts will be selected are asymptomatic adults from the urban areas of Berlin, Cologne, Frankfurt (Main), Hamburg, and Munich with no history of heart failure who have one or more risk factor for developing heart failure. They are either volunteers or referred from local cardiologists.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2025-09-13 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of asymptomatic pre-heart failure (stage B) in an urban population | at baseline
  Asymptomatic pre-heart failure (stage B) is defined as CMR-derived global longitudinal strain (GLS) ≥ -15%

SECONDARY OUTCOMES:
Prevalence of chronic kidney disease (CKD) | at baseline
  CKD is defined as eGFR < 60%
Adherence to therapy | 5 years and 10 years later
  Assessed using the MARS-10 questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sebastian Kelle, Prof. Dr., Principal Investigator — Deutsches Herzzentrum der Charité
Locations (1):
- Deutsches Herzzentrum der Charité, Berlin, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] NVL Chronische Herzinsuffizienz Langfassung - Version 4.0, 2023
- [Background] Spertus JA, Jones PG, Sandhu AT, Arnold SV. Interpreting the Kansas City Cardiomyopathy Questionnaire in Clinical Trials and Clinical Care: JACC State-of-the-Art Review. J Am Coll Cardiol. 2020 Nov 17;76(20):2379-2390. doi: 10.1016/j.jacc.2020.09.542. PMID 33183512
- [Background] Leotsinidis M, Alexopoulos A, Schinas V, Kardara M, Kondakis X. Plasma retinol and tocopherol levels in greek elderly population from an urban and a rural area: associations with the dietary habits. Eur J Epidemiol. 2000;16(11):1009-16. doi: 10.1023/a:1010895227352. PMID 11421468
- [Background] Cuetara MS, del Palacio A, Pereiro M, Amor E, Alvarez C, Noriega AR. Prevalence of undetected tinea capitis in a school survey in Spain. Mycoses. 1997 Sep;40(3-4):131-7. doi: 10.1111/j.1439-0507.1997.tb00202.x. PMID 9375502
- [Background] Brooks EG, Klimpel GR, Vaidya SE, Keeney SE, Raimer S, Goldman AS, Schmalstieg FC. Thymic hypoplasia and T-cell deficiency in ectodermal dysplasia: case report and review of the literature. Clin Immunol Immunopathol. 1994 Apr;71(1):44-52. doi: 10.1006/clin.1994.1050. PMID 8137558
- [Background] Yang H, Negishi K, Wang Y, Nolan M, Marwick TH. Imaging-Guided Cardioprotective Treatment in a Community Elderly Population of Stage B Heart Failure. JACC Cardiovasc Imaging. 2017 Mar;10(3):217-226. doi: 10.1016/j.jcmg.2016.11.015. PMID 28279368
- [Background] Whitmore K, Zhou Z, Chapman N, Huynh Q, Magnussen CG, Sharman JE, Marwick TH. Impact of Patient Visualization of Cardiovascular Images on Modification of Cardiovascular Risk Factors: Systematic Review and Meta-Analysis. JACC Cardiovasc Imaging. 2023 Aug;16(8):1069-1081. doi: 10.1016/j.jcmg.2023.03.007. Epub 2023 May 24. PMID 37227327
- [Background] Renton AM, Whitaker L, Riddlesdell M. Heterosexual HIV transmission and STD prevalence: predictions of a theoretical model. Sex Transm Infect. 1998 Oct;74(5):339-44. doi: 10.1136/sti.74.5.339. PMID 10195029
- [Background] Hood SR, Giazzon AJ, Seamon G, Lane KA, Wang J, Eckert GJ, Tu W, Murray MD. Association Between Medication Adherence and the Outcomes of Heart Failure. Pharmacotherapy. 2018 May;38(5):539-545. doi: 10.1002/phar.2107. Epub 2018 Apr 30. PMID 29600819
- [Background] Patchell RA, Posner JB. Neurologic complications of systemic cancer. Neurol Clin. 1985 Nov;3(4):729-50. PMID 3908895
- [Background] Bozkurt B, Ahmad T, Alexander KM, Baker WL, Bosak K, Breathett K, Fonarow GC, Heidenreich P, Ho JE, Hsich E, Ibrahim NE, Jones LM, Khan SS, Khazanie P, Koelling T, Krumholz HM, Khush KK, Lee C, Morris AA, Page RL 2nd, Pandey A, Piano MR, Stehlik J, Stevenson LW, Teerlink JR, Vaduganathan M, Ziaeian B; Writing Committee Members. Heart Failure Epidemiology and Outcomes Statistics: A Report of the Heart Failure Society of America. J Card Fail. 2023 Oct;29(10):1412-1451. doi: 10.1016/j.cardfail.2023.07.006. Epub 2023 Sep 26. No abstract available. PMID 37797885
- [Background] Haji K, Huynh Q, Wong C, Stewart S, Carrington M, Marwick TH. Improving the Characterization of Stage A and B Heart Failure by Adding Global Longitudinal Strain. JACC Cardiovasc Imaging. 2022 Aug;15(8):1380-1387. doi: 10.1016/j.jcmg.2022.03.007. Epub 2022 May 11. PMID 35926896
- [Background] Potter E, Stephenson G, Harris J, Wright L, Marwick TH. Screening-guided spironolactone treatment of subclinical left ventricular dysfunction for heart failure prevention in at-risk patients. Eur J Heart Fail. 2022 Apr;24(4):620-630. doi: 10.1002/ejhf.2428. Epub 2022 Jan 27. PMID 35014128
- [Background] Chistoni GC. [Some problems posed by double-blind investigation of psychotropic drugs: clinical trial of Nobrium Roche]. Schweiz Arch Neurol Neurochir Psychiatr. 1971;108(2):309-15. No abstract available. French. PMID 4941608
- [Background] Komajda M, Cowie MR, Tavazzi L, Ponikowski P, Anker SD, Filippatos GS; QUALIFY Investigators. Physicians' guideline adherence is associated with better prognosis in outpatients with heart failure with reduced ejection fraction: the QUALIFY international registry. Eur J Heart Fail. 2017 Nov;19(11):1414-1423. doi: 10.1002/ejhf.887. Epub 2017 Apr 30. PMID 28463464
- See also: Datenbank der Gesundheitsberichterstattung (GBE) der Länder — http://www.gbe-bund.de
- See also: NHS Diagnostic Waiting Times and Activity Statistical Report — https://www.england.nhs.uk/statistics/wp-content/uploads/sites/2/2024/01/DWTA-Report-November-2023_8HO7S.pdf